CLINICAL TRIAL: NCT02586207
Title: Phase Ib Study of Pembrolizumab in Combination With Chemo Radiotherapy (CRT) for Locally-advanced Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Pembrolizumab in Combination With CRT for LA-SCCHN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanford Health (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SH MISP203
Record Dates: First submitted 2015-10-20; First posted 2015-10-26 (Estimated); Results first posted 2021-01-15 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Cancer; Squamous Cell Carcinoma; Oral Cavity Cancer; Oropharynx Cancer; Hypopharynx Cancer; Larynx Cancer; Laryngeal Cancer
Keywords: Larynx; Squamous Cell; Oral cavity; Oropharynx; Hypopharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell; Mouth Neoplasms; Oropharyngeal Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Laryngeal Diseases | interventions — pembrolizumab; Cisplatin; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): Pembrolizumab + Cisplatin + Radiation
  Interventions: Drug: pembrolizumab (MK-3475); Drug: Cisplatin; Radiation: Radiation

INTERVENTIONS:
Drug: pembrolizumab (MK-3475) — 200mg IV on days -7(loading dose), 15, 36, 57, 78, 99, 120, 141.
  Other Names: Keytruda
Drug: Cisplatin — Cisplatin 40 mg/m2 IV on days 1, 8, 15, 22, 29, 36
  Other Names: Platinol, Platinol-AQ
Radiation: Radiation — 70 Gy fractionated over 35 days

SUMMARY:
This is a single-arm, multi-site, open-label trial of pembrolizumab (MK-3475) used in combination with standard, cisplatin-based, definitive chemoradiotherapy (CRT) in patients with stage III-IVB squamous cell carcinoma of the head and neck (SCCHN). Approximately 39 patients with Stage III-IVB SCCHN will be enrolled to evaluate both the safety and efficacy of this novel combination. Subjects will not be randomized and will all receive the study treatment.

Treatment will consist of a loading dose of pembrolizumab 200 mg IV given 7 days prior to initiation of CRT (day-7). CRT with cisplatin 40 mg/m2 IV weekly and head and neck radiation at 70 Gy fractionated at 2 Gy once daily over 35 days, will begin on day 1. CRT will end on approximately day 46-50. Pembrolizumab 200 mg IV will continue following CRT in an adjuvant fashion starting on day 57 for an additional 5 doses, as tolerated, through day 141. Subjects will be evaluated for response following treatment.

DETAILED DESCRIPTION:
Each subject will participate in the trial from the time the subject signs the Informed Consent Form (ICF) through the final protocol-specified contact. After a screening phase of 28 days, eligible subjects will receive treatment on Day -7 with a loading dose of the study drug. This will continue during concurrent therapy with cisplatin and radiation, which will begin on day 1. Treatment will continue until completion of therapy, documented confirmed disease progression, unacceptable adverse event(s), intercurrent illness that prevents further administration of treatment, investigator's decision to withdraw the subject, subject withdraws consent, pregnancy of the patient, noncompliance with trial treatment or procedure requirements; or administrative reasons. After the end of treatment, each patient will be followed for 30 days for adverse event monitoring (serious adverse events will be collected for 90 days after the end of treatment or 30 days after the end of treatment if the patient initiates new anticancer therapy, whichever is earlier). Subjects who discontinue for reasons other than disease progression will have post-treatment follow-up for disease status until end of study disease progression, initiating a non-study cancer treatment, withdrawing consent, or becoming lost to follow-up. All subjects will be followed by telephone for overall survival until death, withdrawal of consent, or the Investigator is notified by Sanford Research to discontinue follow-up

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically or cytologically-confirmed head and neck squamous cell carcinoma of the oral cavity (excluding lip), oropharynx, hypopharynx, or larynx.
2. Have TNM clinical stage III, IVA, or IVB disease
3. Be eligible for curative-intent concurrent chemoradiation therapy
4. Be willing and able to provide written informed consent for the trial.
5. Be 18 years of age on day of signing informed consent.
6. Have measurable disease based on RECIST 1.1.
7. Be willing to provide tissue from a recently obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day -7. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from Sanford Research.
8. Have a performance status of 0 or 1 on the ECOG Performance Scale.
9. Demonstrate adequate organ function as defined:

   Absolute neutrophil count (ANC) ≥1,500 /mcL Platelets ≥100,000 / mcL Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment) Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases Albumin >2.5 mg/dL
10. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
11. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
12. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Patients may not be receiving any other investigational agents, chemotherapy, immunotherapy, radiotherapy, or molecular targeted agents within 4 weeks of the start of the study treatment.
2. Prior treatment with radiation to the head and neck
3. Patients with TNM Stage IVC disease
4. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
5. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
6. Has a known history of active TB (Bacillus Tuberculosis)
7. Hypersensitivity to pembrolizumab or any of its excipients.
8. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
9. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy.
10. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
11. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
12. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
13. Has known history of, or any evidence of active, non-infectious pneumonitis.
14. Has an active infection requiring systemic therapy.
15. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
16. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
17. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120days after the last dose of trial treatment.
18. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
19. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
20. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
21. Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-11; Primary Completion 2020-09-29 (Actual); Study Completion 2025-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven F Powell, MD, Principal Investigator — Sanford Research
Locations (4):
- United States (4):
  - UCSD Moores Cancer Center, La Jolla, California
  - Sanford-Bismarck Medical Center, Bismarck, North Dakota
  - Sanford-Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Health Cancer Center, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: Yes
Projected to share initial safety data 4th quarter 2016

REFERENCES:
- [Background] Spanos WC, Nowicki P, Lee DW, Hoover A, Hostager B, Gupta A, Anderson ME, Lee JH. Immune response during therapy with cisplatin or radiation for human papillomavirus-related head and neck cancer. Arch Otolaryngol Head Neck Surg. 2009 Nov;135(11):1137-46. doi: 10.1001/archoto.2009.159. PMID 19917928
- [Background] Vermeer DW, Spanos WC, Vermeer PD, Bruns AM, Lee KM, Lee JH. Radiation-induced loss of cell surface CD47 enhances immune-mediated clearance of human papillomavirus-positive cancer. Int J Cancer. 2013 Jul;133(1):120-9. doi: 10.1002/ijc.28015. Epub 2013 Feb 12. PMID 23292955
- [Background] Lyford-Pike S, Peng S, Young GD, Taube JM, Westra WH, Akpeng B, Bruno TC, Richmon JD, Wang H, Bishop JA, Chen L, Drake CG, Topalian SL, Pardoll DM, Pai SI. Evidence for a role of the PD-1:PD-L1 pathway in immune resistance of HPV-associated head and neck squamous cell carcinoma. Cancer Res. 2013 Mar 15;73(6):1733-41. doi: 10.1158/0008-5472.CAN-12-2384. Epub 2013 Jan 3. PMID 23288508
- [Background] Seiwert T, Burtness B, Weiss J, Gluck I, Eder JP, Pai SI, et al. A phase IB study of MK-3475 in patients with human papilloma virus (HPV) associated and non-HPV associated head and neck (H/N) cancer. ASCO 2014 Abstract #6011, Jun 2014.
- [Background] Dovedi SJ, Adlard AL, Lipowska-Bhalla G, McKenna C, Jones S, Cheadle EJ, Stratford IJ, Poon E, Morrow M, Stewart R, Jones H, Wilkinson RW, Honeychurch J, Illidge TM. Acquired resistance to fractionated radiotherapy can be overcome by concurrent PD-L1 blockade. Cancer Res. 2014 Oct 1;74(19):5458-68. doi: 10.1158/0008-5472.CAN-14-1258. PMID 25274032
- [Background] Parikh F, Duluc D, Imai N, Clark A, Misiukiewicz K, Bonomi M, Gupta V, Patsias A, Parides M, Demicco EG, Zhang DY, Kim-Schulze S, Kao J, Gnjatic S, Oh S, Posner MR, Sikora AG. Chemoradiotherapy-induced upregulation of PD-1 antagonizes immunity to HPV-related oropharyngeal cancer. Cancer Res. 2014 Dec 15;74(24):7205-16. doi: 10.1158/0008-5472.CAN-14-1913. Epub 2014 Oct 15. PMID 25320012
- [Derived] Powell SF, Gold KA, Gitau MM, Sumey CJ, Lohr MM, McGraw SC, Nowak RK, Jensen AW, Blanchard MJ, Fischer CD, Bykowski J, Ellison CA, Black LJ, Thompson PA, Callejas-Valera JL, Lee JH, Cohen EEW, Spanos WC. Safety and Efficacy of Pembrolizumab With Chemoradiotherapy in Locally Advanced Head and Neck Squamous Cell Carcinoma: A Phase IB Study. J Clin Oncol. 2020 Jul 20;38(21):2427-2437. doi: 10.1200/JCO.19.03156. Epub 2020 Jun 1. PMID 32479189

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm
Started | 59
Completed | 57
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 59
Age, Continuous [Median (Full Range); unit: years] | 59.8 [36 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 58
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 57
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events Will be Assessed and Graded Using CTCAE 4.0. Occurrences With Max Grade and Percentage/Number of Participants Affected by AEs Will be Provided.
Description: To determine the safety and tolerability of pembrolizumab given in combination with cisplatin-based chemoradiotherapy (CRT) in subjects with treatment naive Stage III-IVB squamous cell carcinoma of the head and neck (SCCHN).
  Number of participants affected by AEs will be reported by grade and percentage of participants affected.
  Safety and tolerability will be assessed by clinical review of all relevant parameters including adverse events (AEs), laboratory tests, and vital signs. Count and percentage of AE will be provided.
Time Frame: through day 240 (this time frame allows capturing of AEs that occurred up to 90 days after completion of treatment)
Population: Number of participants who experience an Adverse Event.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 57
Participants | 57

2. Secondary Outcome: Evaluation of the Efficacy of Pembrolizumab Given in Combination With Definitive CRT by Determining the Number of Participants With Complete Response at Treatment End (Day 150)
Description: Response was determined using a composite end point of overall end-of-treatment (EOT) complete response (CR) at day 150 (approximately 12 weeks after completion of chemoradiotherapy) by CT of the neck (RECIST 1.1).
  Optional positron emission tomography (PET) imaging was allowed rather than neck dissection if CT could not confirm CR. Complete metabolic response was assessed using Hopkins score of 1, 2, or 3 on PET imaging. For those without an imaging CR, pathologic confirmation was recommend (but not required) by selective neck dissection and/or directed biopsy of the suspected active disease site. If pathologic evaluation of the potential disease site confirmed no residual invasive or in situ cancer, the patient was determined to have a pathologic CR. In cases with both an imaging CR and pathologic response assessment, the pathologic response defined final overall response. Therefore, patients with a final EOT CR included those with either an imaging (CT or PET) or pathologic CR.
Time Frame: Day 150 (post treatment imaging)
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 57
Participants | 47

ADVERSE EVENTS:
Time Frame: Enrollment through Day 150 plus 90 days for SAE reporting
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 10/59
Serious Adverse Events (participants affected / at risk) | 28/59
Other Adverse Events (participants affected / at risk) | 59/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=59)
Adrenal Insufficiency (Endocrine disorders) | 1
Aspiratoin Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3
cardiac arrest (Cardiac disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 7
Dysphagia (Gastrointestinal disorders) | 4
Encephalitis Infection (Infections and infestations) | 1
Fever (General disorders) | 3
Gastric Ulcer (Gastrointestinal disorders) | 1
GI Bleed (Gastrointestinal disorders) | 1
Hyponatrimia (Metabolism and nutrition disorders) | 2
Ileus (Gastrointestinal disorders) | 1
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 2
Lowet gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Neoplasms benign, malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neutropenic Fever (Blood and lymphatic system disorders) | 1
Pain (General disorders) | 2
Palpitations (Cardiac disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Sepsis (Infections and infestations) | 1
Syncope (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Urinary Tract Infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 3
Weight Loss (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=59)
Lymphocyte Count Decreased (Investigations) | 58
Anemia (Blood and lymphatic system disorders) | 56
White Blood Cell Decreased (Investigations) | 55
Dysphagia (Gastrointestinal disorders) | 51
Weight Loss (Investigations) | 50
Dermatitis radiation (Injury, poisoning and procedural complications) | 52
Dry Mouth (Gastrointestinal disorders) | 50
Fatigue (General disorders) | 51
Nausea (Gastrointestinal disorders) | 48
Mucositis oral (Gastrointestinal disorders) | 48
Dysgeusia (Nervous system disorders) | 47
Hyponatremia (Metabolism and nutrition disorders) | 45
Constipation (Gastrointestinal disorders) | 41
Salivary Duct Inflammation (Gastrointestinal disorders) | 41
neutrophil count decreased (Investigations) | 39
Vomiting (Gastrointestinal disorders) | 35
Hypomagnesemia (Metabolism and nutrition disorders) | 36
Anorexia (Metabolism and nutrition disorders) | 34
Platelet count decreased (Investigations) | 34
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 33
Abdominal Pain (Gastrointestinal disorders) | 4
Alanine aminotransferase increased (Investigations) | 14
Alkaline phosphatase increased (Investigations) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 15
Anxiety (Psychiatric disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Aspartate aminotransferase increased (Investigations) | 10
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 7
Ear pain (Ear and labyrinth disorders) | 8
Hearing impaired (Ear and labyrinth disorders) | 9
Tinnitus (Ear and labyrinth disorders) | 19
Blurred vision (Eye disorders) | 4
Dry Eye (Eye disorders) | 3
Hyperthyroidism (Endocrine disorders) | 10
Hypothyroidism (Endocrine disorders) | 21
Chills (General disorders) | 11
Colitis (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 29
Dyspepsia (Gastrointestinal disorders) | 8
Edema Limbs (General disorders) | 8
Fever (General disorders) | 9
Flu like symptoms (General disorders) | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 6
Malaise (General disorders) | 5
Neck edema (General disorders) | 6
Oral pain (Gastrointestinal disorders) | 16
pain (General disorders) | 19
Fall (Injury, poisoning and procedural complications) | 7
Infections and infestations - Other, specify (Infections and infestations) | 3
Mucosal infection (Infections and infestations) | 19
Skin Infection (Infections and infestations) | 6
Blood bilirubin increased (Investigations) | 3
Creatinine increased (Investigations) | 9
Lymphocyte count increased (Investigations) | 9
Dehydration (Metabolism and nutrition disorders) | 29
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 6
Hypermagnesemia (Metabolism and nutrition disorders) | 3
Hyperuricemia (Metabolism and nutrition disorders) | 13
Hypoalbuminemia (Metabolism and nutrition disorders) | 23
Hypocalcemia (Metabolism and nutrition disorders) | 13
Hypokalemia (Metabolism and nutrition disorders) | 21
Hypophosphatemia (Metabolism and nutrition disorders) | 15
Back pain (Musculoskeletal and connective tissue disorders) | 5
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Trismus (Musculoskeletal and connective tissue disorders) | 9
Headache (Nervous system disorders) | 13
Paresthesia (Nervous system disorders) | 3
Peripheral motor neuropathy (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 14
Syncope (Nervous system disorders) | 3
Confusion (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 11
Insomnia (Psychiatric disorders) | 17
Hematuria (Renal and urinary disorders) | 11
Proteinuria (Renal and urinary disorders) | 21
Urinary frequency (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 17
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 9
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 23
Rash acneiform (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 12
Hot flashes (Vascular disorders) | 4
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 14
Lymphedema (Vascular disorders) | 25
Dizziness (Nervous system disorders) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/07/NCT02586207/Prot_SAP_000.pdf